CLINICAL TRIAL: NCT06813391
Title: Prevalence of Central Neuropathic Pain After a Stroke in Patients Attending Post-stroke Consultations in the Île-de-France Region
Acronym: AVCD
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: AVCD
Record Dates: First submitted 2025-01-30; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Stroke Sequelae; Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Patient Reported Outcome (PRO) — after enrollment, patient will answer to several PRO to assess their pain and overall well-being after their stroke

SUMMARY:
Post-stroke pain is common, affecting 15-50% of patients and significantly impacting their quality of life, rehabilitation, and functional recovery. There are different types of post-stroke pain, including peripheral pain related to spasticity, shoulder pain, complex regional pain syndrome, and headaches, as well as central pain linked to brain lesions. Central Post-Stroke Pain (CPSP) is diagnosed when the pain has neuropathic characteristics (burning, cold, tightness, compression), possibly accompanied by allodynia, hyperesthesia, and sensory-motor disorders localized to the area affected by the stroke. CPSP disrupts sleep, impairs functional rehabilitation, and can lead to depression, anxiety, substance abuse, and cognitive disorders. The prevalence of CPSP varies, ranging from 1% to 35%, but it is likely underreported due to difficulties in detection caused by cognitive or communication issues, the clinical variability of CPSP, and its coexistence with other types of post-stroke pain.

CPSP often remains resistant to standard neuropathic pain treatments, such as anticonvulsants and antidepressants, which may cause side effects that reduce patients' autonomy and quality of life. Non-pharmacological therapies used in other chronic pain conditions may offer promising alternatives, but have not been widely studied in CPSP. Improved clinical characterization of CPSP patients is essential. Following a 2015 decree by the French Ministry of Health, post-stroke consultations are standardized, providing a good opportunity for systematic pain screening. The study proposes a systematic screening of different types of pain during post-stroke consultations, categorizing patients into three groups: those with CPSP, those with pain from another mechanism, and those without pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥18 years
* Patient attending a post-stroke consultation (3 to 6 months after the stroke)
* Stroke confirmed by imaging (MRI or CT scan)
* Francophone patient
* Patient not opposing participation in the study

Exclusion Criteria:

* Patient with cognitive or communication disorders preventing them from completing the questionnaires (as assessed by the investigator)
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post Stroke Patient
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Central Pain | enrollment
  determine the prevalence of post-stroke central pain in patients recruited during post-stroke consultations conducted between 3 and 6 months after their stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Paris Saint Joseph, Paris, France, France

IPD SHARING:
Plan to Share IPD: No